CLINICAL TRIAL: NCT05604612
Title: Assessment of the Effectiveness of Corticision Combined by Selfligating Bracket System on the Acceleration of Orthodontic Tooth Movement; A Prospective Clinical Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Hazem Abd Elhafeez Abd Elkhalek, Hazem Abd Elhafeez, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 721/271
Record Dates: First submitted 2022-10-30; First posted 2022-11-03 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Orthodontic Appliance Complication

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental)
  Interventions: Procedure: Corticision
- Active Comparator (No Intervention)

INTERVENTIONS:
Procedure: Corticision — Incisions in the cortical plate of maxillary bone
  Arms: Experimental

SUMMARY:
the goal of this clinical trial is to assess the effectiveness of the corticision with self-ligating bracket system on the acceleration of orthodontic tooth movement.The main question it aims to answer is whether or not there would be an augmented effect by undergoing corticision with using self-ligating brackets regarding the acceleration of orthodontic tooth movement.

ELIGIBILITY:
Inclusion Criteria:

* Class I orthodontic patients with mild to moderate crowding of upper anterior segment (2-4 mm) All permanent teeth are erupted (3rd molar not included). Good oral and general health No systemic disease or regular medication that could interfere and/or affect orthodontic teeth movement No previous orthodontic treatment.

Exclusion Criteria:

* Orthodontic cases with severe crowding of upper anterior segment that require extraction treatment approach. Patients with a blocked-out tooth that will not allow for placement of the bracket at the initial bonding appointment. Patients with untreated decay or endodontic lesion.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 16 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Little's Irregularity Index | two months
  crowding resolution